CLINICAL TRIAL: NCT01446809
Title: The Effect of Antiangiogenic Therapy With Pazopanib Prior to Preoperative Chemotherapy for Subjects With Extremity Soft Tissue Sarcomas: A Randomized Study to Evaluate Response by Imaging
Brief Title: Pazopanib Hydrochloride Followed by Chemotherapy and Surgery in Treating Patients With Soft Tissue Sarcoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 7487; NCI-2011-02488 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 7487 (Other: Fred Hutch/University of Washington Cancer Consortium); P30CA015704 (NIH)
Record Dates: First submitted 2011-09-12; First posted 2011-10-05 (Estimated); Results first posted 2019-04-25 (Actual); Last update posted 2020-04-13 (Actual); Status verified 2020-01

CONDITIONS: Stage IIA Adult Soft Tissue Sarcoma; Stage III Adult Soft Tissue Sarcoma; Stage IV Adult Soft Tissue Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — Doxorubicin; Ifosfamide; pazopanib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (pazopanib hydrochloride) (Experimental): Patients receive pazopanib hydrochloride PO QD. Treatment continues for 14 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Doxorubicin Hydrochloride; Radiation: External Beam Radiation Therapy; Drug: Ifosfamide; Other: Laboratory Biomarker Analysis; Drug: Pazopanib Hydrochloride; Other: Pharmacological Study; Procedure: Therapeutic Conventional Surgery
- Arm II (placebo) (Placebo Comparator): Patients receive placebo PO QD. Treatment continues for 14 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Doxorubicin Hydrochloride; Radiation: External Beam Radiation Therapy; Drug: Ifosfamide; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Other: Placebo; Procedure: Therapeutic Conventional Surgery

INTERVENTIONS:
Drug: Doxorubicin Hydrochloride — Given IV
  Other Names: 5,12-Naphthacenedione, 10-[(3-amino-2,3,6-trideoxy-alpha-L-lyxo-hexopyranosyl)oxy]-7,8, 9,10-tetrahydro-6,8,11-trihydroxy-8-(hydroxyacetyl)-1-methoxy-, hydrochloride, (8S-cis)- (9CI); ADM; Adriacin; Adriamycin; Adriamycin Hydrochloride; Adriamycin PFS; Adriamycin RDF; ADRIAMYCIN, HYDROCHLORIDE; Adriamycine; Adriblastina; Adriblastine; Adrimedac; Chloridrato de Doxorrubicina; DOX; DOXO-CELL; Doxolem; Doxorubicin.HCl; Doxorubin; Farmiblastina; FI 106; FI-106; hydroxydaunorubicin; Rubex
Radiation: External Beam Radiation Therapy — Undergo external beam radiation therapy
  Other Names: Definitive Radiation Therapy; EBRT; External Beam Radiotherapy; External Beam RT; external radiation; External Radiation Therapy; external-beam radiation
Drug: Ifosfamide — Given IV
  Other Names: Asta Z 4942; Asta Z-4942; Cyfos; Holoxan; Holoxane; Ifex; IFO; IFO-Cell; Ifolem; Ifomida; Ifomide; Ifosfamidum; Ifoxan; IFX; Iphosphamid; Iphosphamide; Iso-Endoxan; Isoendoxan; Isophosphamide; Mitoxana; MJF 9325; MJF-9325; Naxamide; Seromida; Tronoxal; Z 4942; Z-4942
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Pazopanib Hydrochloride — Given PO
  Other Names: GW786034B; Votrient
  Arms: Arm I (pazopanib hydrochloride)
Other: Pharmacological Study — Correlative studies
Other: Placebo — Given PO
  Other Names: placebo therapy; PLCB; sham therapy
  Arms: Arm II (placebo)
Procedure: Therapeutic Conventional Surgery — Undergo surgery

SUMMARY:
This randomized pilot clinical trial studies pazopanib hydrochloride followed by chemotherapy and surgery in treating patients with soft tissue sarcoma. Pazopanib hydrochloride may stop the growth of tumor cells by blocking some of the enzymes that are needed for cell growth and may also stop the growth of soft tissue sarcoma by blocking blood flow to the tumor. Giving pazopanib hydrochloride and chemotherapy before surgery may make the tumor smaller and reduce the amount of tissue that needs to be removed.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the absolute values and changes in standardized uptake values (SUV) by fludeoxyglucose F18 (FDG)-positron emission tomography (PET) before and after a 14 day Run-in period of pazopanib (pazopanib hydrochloride) versus placebo, and to compare this to the change in SUV following pre-operative chemotherapy.

II. To evaluate the correlation between antiangiogenic activity and pazopanib drug exposure.

III. To assess the response rate by Response Evaluation Criteria In Solid Tumors (RECIST) criteria after the 14 day Run-in period of pazopanib versus placebo and compare this to the response rate following pre-operative chemotherapy.

SECONDARY OBJECTIVES:

I. To examine the activity of antiangiogenic therapy with pazopanib combined with pre-operative chemotherapy for high risk extremity soft tissue sarcomas as measured by: histological necrosis at surgery; change in plasma and tumor biomarker assays of angiogenesis

II. To evaluate the safety of sequential treatment with pazopanib and pre-operative chemotherapy with doxorubicin (doxorubicin hydrochloride) and ifosfamide.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive pazopanib hydrochloride orally (PO) once daily (QD). Treatment continues for 14 days in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive placebo PO QD. Treatment continues for 14 days in the absence of disease progression or unacceptable toxicity.

All patients then receive neoadjuvant chemotherapy comprising doxorubicin hydrochloride intravenously (IV) continuously over days 1-3 and ifosfamide IV on days 1-5. Treatment repeats every 21 days for 4 courses. Beginning 2-4 weeks later, all patients undergo surgery followed by 2 more courses of chemotherapy 2-4 weeks after completion of surgery. Some patients may also undergo adjuvant external beam radiation therapy 5 days a week for 5 days followed by a boost. Patients treated on Arm I may resume pazopanib hydrochloride 1 week after completion of all adjuvant therapy for up to 1 year. Treatment continues in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed soft-tissue sarcoma, excluding alveolar and embryonal rhabdomyosarcoma, well- and dedifferentiated adipocytic sarcomas, Ewing's, osteosarcoma, or gastrointestinal stromal tumor; American Joint Committee on Cancer (AJCC) (6th Edition) Stage III or T2a Stage II or Stage IV treatment naive patients planned for resection of the primary tumor, with resectable metastatic disease
* Measurable disease greater than 5 centimeters in greatest dimension; measurable lesions are defined as those that can be accurately measured in at least one dimension (longest diameter for non-nodal lesions and short axis for nodal lesions to be recorded) by chest x-ray, computed tomography (CT) scan, magnetic resonance imaging (MRI) or with calipers by clinical exam; all tumor measurements must be recorded in millimeters (or decimal fractions of centimeters)
* Intermediate or high grade lesions: 2 or 3 on a scale of 1-3 or grades 2 to 4 on a scale of 1-4
* Sarcoma located on upper (includes shoulder) or lower (includes hip) extremities or on the body wall
* Life expectancy of greater than 6 months
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1
* Karnofsky >= 80%
* No prior chemotherapy, radiotherapy, or antiangiogenic therapy
* Absolute neutrophil count (ANC) >= 1500/uL
* Hemoglobin (Hgb) >= 9.0 g/dL
* Platelets >= 100,000/uL
* Creatinine =< 1.5 x upper limit of normal (ULN)
* Bilirubin =< 1.5 mg/dL
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) =< 1.5 x ULN
* Prothrombin time (PT)/international normalized ratio (INR)/partial thromboplastin time (PTT) within 1.2 X the ULN unless a subject is receiving Coumadin and has stable INR which is in range for the desired level of anticoagulation
* Left ventricular ejection fraction (LVEF) >= 50%
* Blood pressure (BP) no greater than 140 mmHg (systolic) and 90 mmHg (diastolic) for eligibility; initiation or adjustment of BP medication is permitted prior to study entry provided that the average of three BP readings on baseline assessment prior to enrollment is less than 140/90 mmHg
* Eligibility of subjects receiving any medications or substances known to affect or with the potential to affect the activity or pharmacokinetics of pazopanib will be determined following review of their cases by the Principal Investigator
* Women of child-bearing potential and men must agree to use adequate contraception
* A female is eligible to enter and participate in this study if she is of non-childbearing potential (i.e., physiologically incapable of becoming pregnant) or if she is of childbearing potential
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Subjects with known brain metastases and/or unresectable sarcoma
* Uncontrolled intercurrent illness including, active serious infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac ventricular arrhythmia requiring anti-arrhythmic therapy, serious hepatic impairment, or psychiatric illness/social situations that would limit compliance with study
* Pregnant or lactating women
* Subjects with no additional active malignancy within the last 3 years
* Subjects receiving other investigational agents
* Subjects with a history of allergic reactions attributed to compounds of similar chemical or biologic composition to pazopanib or other agents used in the study
* Subjects who have both bilirubin > ULN and AST/ALT > ULN
* Subjects with a urine protein/creatinine ratio greater than 1
* Subjects with a baseline corrected QT (QTc) of equal to or greater than 480 msecs or other significant electrocardiogram (ECG) abnormalities
* Certain medications that act through the cytochrome P450 (CYP450) system are specifically prohibited in subjects receiving pazopanib and others should be avoided or administered with extreme caution and require principal investigator (PI) approval

  * Strong inhibitors of CYP3A4 such as ketoconazole, itraconazole, clarithromycin, atazanavir, indinavir, nefazodone, nelfinavir, ritonavir, saquinavir, telithromycin, voriconazole may increase pazopanib concentrations and are prohibited; grapefruit juice is also an inhibitor of CYP450 and should not be taken with pazopanib
  * Strong inducers of CYP3A4, such as rifampin, may decrease pazopanib concentrations, are prohibited
  * Medications which have narrow therapeutic windows and are substrates of CYP3A4, CYP2D6, or CYP2C8 should be avoided and, if necessary, administered with caution
  * Pazopanib, 800 mg once daily, has no effect on CYP2C9, CYP1A2, or CYP2C19 in vivo but does in vitro; therefore, therapeutic doses of warfarin, a substrate of CYP2C9, and omeprazole, a substrate of CYP2C19 are permitted; caffeine, a substrate of CYP1A2, is also permitted
* Certain medications that are associated with a risk for QTc prolongation and/or Torsades de Pointes, although not prohibited, should be avoided or replaced with medications that do not carry these risks, if possible
* Subjects who require heparin other than low-molecular weight heparin
* Subjects with any condition that may impair the ability to swallow or absorb oral medications/investigational product including:

  * Any lesion, whether induced by tumor, radiation or other conditions, which makes it difficult to swallow capsules or pills
  * Prior surgical procedures affecting absorption including, but not limited to major resection of stomach or small bowel
  * Active peptic ulcer disease, not on a proton pump inhibitor
  * Malabsorption syndrome
* Subjects with any condition that may increase the risk of gastrointestinal bleeding or gastrointestinal perforation, including

  * Active peptic ulcer disease, not on a proton pump inhibitor
  * Known intraluminal metastatic lesions
  * Inflammatory bowel disease (e.g., ulcerative colitis, Crohn's disease) or
  * Other gastrointestinal conditions which increase the risk of perforation
  * History of abdominal fistula, gastrointestinal perforation or intra-abdominal abscess within 28 days prior to beginning study treatment
* Subjects with any of the following cardiovascular conditions within the past 6 months:

  * Cerebrovascular accident (CVA) or transient ischemic attack (TIA)
  * Cardiac arrhythmia
  * Admission for unstable angina
  * Cardiac angioplasty or stenting
  * Coronary artery bypass graft surgery
  * Pulmonary embolism, untreated deep venous thrombosis (DVT) or DVT which has been treated with therapeutic anticoagulation for less than 6 weeks
  * Arterial thrombosis
  * Symptomatic peripheral vascular disease
  * Class III or IV heart failure as defined by the New York Heart Association (NYHA) functional classification system; a subject who has a history of Class II heart failure and is asymptomatic on treatment may be considered eligible
* History of hemoptysis in excess of 2.5 mL (1/2 teaspoon ) within 8 weeks prior to first dose of study drug
* History of serious or non-healing wound, ulcer, or bone fracture
* Human immunodeficiency virus (HIV)-positive subjects on combination antiretroviral therapy are ineligible
* Subjects with severe hepatic impairment

  * Bilirubin > 3 x ULN, regardless of any level of ALT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2012-04; Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Darin Davidson, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Pazopanib: Patients receive pazopanib hydrochloride PO QD. Treatment continues for 14 days in the absence of disease progression or unacceptable toxicity.
  Doxorubicin Hydrochloride: Given IV External Beam Radiation Therapy: Undergo external beam radiation therapy Ifosfamide: Given IV Laboratory Biomarker Analysis: Correlative studies Pazopanib Hydrochloride: Given PO Pharmacological Study: Correlative studies Therapeutic Conventional Surgery: Undergo surgery
- Placebo: Patients receive placebo PO QD. Treatment continues for 14 days in the absence of disease progression or unacceptable toxicity.
  Doxorubicin Hydrochloride: Given IV External Beam Radiation Therapy: Undergo external beam radiation therapy Ifosfamide: Given IV Laboratory Biomarker Analysis: Correlative studies Pharmacological Study: Correlative studies Placebo: Given PO Therapeutic Conventional Surgery: Undergo surgery
- Blinded: Patients receive pazopanib hydrochloride or placebo PO QD. Patient did not complete study and thus treatment arm remains blinded.
Period: Overall Study
Arm/Group | Pazopanib | Placebo | Blinded
Started | 14 | 7 | 2
Completed | 14 | 7 | 0
Not Completed | 0 | 0 | 2
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Failure to complete study procedures | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pazopanib | Placebo | Total
Number analyzed (Participants) | 14 | 7 | 21
Age, Continuous [Median (Full Range); unit: years] | 49.5 [21 to 70] | 61 [37 to 75] | 53 [21 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 12 | 5 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 13 | 7 | 20
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 13 | 5 | 18
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Screening SUV [Median (Full Range); unit: Standardized Uptake Value- SUV] | 7.1 [2.3 to 38.7] | 9.9 [2.7 to 15.6] | 8.3 [2.3 to 38.7]

OUTCOME MEASURES:

1. Primary Outcome: Change in Maximum SUV of Tumors Measured by FDG-PET Pre- and Post Receipt of Pazopanib Versus Placebo
Description: Change in maximum SUV (standardized uptake value) of tumors measured by FDG-PET. Comparison conducted using a two-sided Wilcoxon rank sum test.
Time Frame: From baseline to 15 days
Measure: Median (Full Range); unit: Standardized uptake value-SUV
Arm/Group | Pazopanib | Placebo
Number analyzed (Participants) | 14 | 7
Standardized uptake value-SUV | -0.1 [-14.7 to 3.5] | -0.1 [-2.2 to 6.0]
Statistical Analysis 1: Comparison: Pazopanib vs Placebo; Test type: Superiority; p = 0.4, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Change in Maximum SUV of Tumors Measured by FDG-PET Post Receipt of 2 Courses of Preoperative Chemotherapy
Description: Change in maximum SUV of tumors measured by FDG-PET. Comparison conducted using a two-sided Wilcoxon rank sum test.
Time Frame: From baseline to 8 weeks
Population: 8 week PET not done on one Pazopanib participant.
Measure: Median (Full Range); unit: SUV
Arm/Group | Pazopanib | Placebo
Number analyzed (Participants) | 13 | 7
SUV | -1.1 [-32.7 to 5.0] | -4.0 [-11.2 to -0.3]
Statistical Analysis 1: Comparison: Pazopanib vs Placebo; Test type: Superiority; p = 0.13, Wilcoxon (Mann-Whitney)

3. Primary Outcome: Tumor Response by RECIST Criteria
Description: RECIST measurements will be performed on serial MRIs to evaluate the correlation with FDG-PET. The longest diameter (LD) of the target lesions will be measured and reported as the baseline LD. The baseline LD will be used as reference to further characterize the objective tumor response of the measurable dimension of the disease.Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Progression (PD), a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: At 15 days
Population: Per RECIST v1.0 for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the LD of target lesions; Progression (PD),20% increase in the sum of the LD of target lesions,or measurable increase in a non-target lesion,or appearance of new lesions.",
Measure: Count of Participants; unit: Participants
Arm/Group | Pazopanib | Placebo
Number analyzed (Participants) | 14 | 7
Participants
  Stable Disease | 14 | 6
  Progressive Disease | 0 | 1

4. Primary Outcome: Tumor Response by RECIST Criteria
Description: as for outcome 3
Time Frame: At 8 weeks
Population: 8 week MRI not done on one Placebo patient.
Measure: Count of Participants; unit: Participants
Arm/Group | Pazopanib | Placebo
Number analyzed (Participants) | 14 | 6
Participants
  Stable Disease | 11 | 5
  Progressive Disease | 2 | 0
  Partial Response | 1 | 1

5. Primary Outcome: Pharmacokinetic Profile of Pazopanib
Description: Trough plasma pazopanib concentration measured during the 14 day run-in period on days 10 through 14.
Time Frame: Up to 14 days
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Pazopanib | Placebo
Number analyzed (Participants) | 14 | 7
ng/mL | 56.38 (0.94) | 0 (0)

6. Secondary Outcome: Change in Levels of VEGF and Soluble VEGFR2 Assessed by ELISA on Plasma and Tumor Extracts
Description: Plasma will be collected for measurement of VEGF and soluble VEGFR2 (sVEGFR2) at baseline, after the 14 day Run-in period of pazopanib, after completion of neoadjuvant chemotherapy and approximately every 3 months thereafter until completion of pazopanib maintenance therapy, when indicated. Quantitative enzyme-linked immunosorbent assays (ELISA) for VEGF and sVEGFR2 will be performed on plasma and tumor extracts. Plasma will also be collected for micro RNA at baseline, after the 14 day Run-in period of pazopanib, following neoadjuvant chemotherapy and every 3 months thereafter until completion of pazopanib maintenance therapy, when indicated.
Time Frame: At baseline and after 14 days
Measure: Number; unit: percentage of concentration
Arm/Group | Pazopanib | Placebo
Number analyzed (Participants) | 14 | 7
percentage of concentration | NA — PI left institution and this data was not analyzed. | NA — PI left institution and this data was not analyzed.

7. Secondary Outcome: Overall Survival
Description: Defined as the interval of time from randomization until death from any cause.
Time Frame: Up to 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Pazopanib | Placebo
Number analyzed (Participants) | 14 | 7
Participants | 12 | 4

8. Secondary Outcome: Number of Participants With Pathologic Response at the Time of Surgery as Measured by % Tumor Viability ( >= 95% Necrosis)
Description: Estimate the amount of viable tumor, and report the percentage of necrosis. Analysis was only completed on a subset of participants.
Time Frame: An expected average of 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Pazopanib | Placebo
Number analyzed (Participants) | 6 | 6
Participants | 6 | 6

9. Secondary Outcome: Progression Free Survival
Description: Defined as the duration of time from randomization to progressive disease (per RECIST), local recurrence, distant metastatic disease (exclusive of stage IV subjects), or death, whichever occurs first.
Time Frame: Up to 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Pazopanib Hydrochloride) | Arm II (Placebo)
Number analyzed (Participants) | 14 | 7
Participants | 10 | 4

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Pazopanib | Placebo | Blinded
All-Cause Mortality (participants affected / at risk) | 2/14 | 3/7 | 2/2
Serious Adverse Events (participants affected / at risk) | 9/14 | 4/7 | 1/2
Other Adverse Events (participants affected / at risk) | 0/14 | 0/7 | 0/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pazopanib (N=14) | Placebo (N=7) | Blinded (N=2)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Tumor Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Febrile Neutropenia (Blood and lymphatic system disorders) | 3 | 4 | 0
Alanine Aminotransferase increased (Investigations) | 1 | 0 | 1
Catheter related infection (Infections and infestations) | 1 | 0 | 0
Platelet count decreased (Investigations) | 4 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1
Mucositis oral (Gastrointestinal disorders) | 1 | 1 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 5 | 0 | 0
Anemia (Blood and lymphatic system disorders) | 2 | 0 | 0
White blood cell decreased (Investigations) | 2 | 1 | 0
Rectal pain (Gastrointestinal disorders) | 1 | 0 | 0
Hypokalemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Bilateral pulmonary emboli (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Endocarditis (Cardiac disorders) | 0 | 0 | 1
Left gluteal abscess (Infections and infestations) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-02): https://cdn.clinicaltrials.gov/large-docs/09/NCT01446809/Prot_SAP_000.pdf